CLINICAL TRIAL: NCT06490367
Title: Safety, Feasibility, and Biomarker Effects of Time-restricted Eating for 12 Weeks in Early-stage Huntington's Disease.
Brief Title: Time-Restricted Eating in Huntington's Disease: A Clinical Pilot Study
Acronym: TREHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Amie Hiller, MD, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00026970
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Huntington Disease
Keywords: Time-restricted eating; Intermittent fasting; Time-restricted feeding; Dietary fasting
MeSH Terms: conditions — Huntington Disease; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Time-Restricted Eating (Experimental): All participants are assigned to this arm.
  Interventions: Behavioral: Time-Restricted Eating Diet

INTERVENTIONS:
Behavioral: Time-Restricted Eating Diet — Participants engage in a time-restricted eating diet, specifically maintaining a 6-8-hour eating window every day for 12 weeks. Participants are allowed to self-select the timing of the eating window, but once selected, they are asked to maintain that schedule daily. Outside of that window, for the remaining 16-18 hours of day/night, participants are asked not to consume calorie-containing food or drink. Beverages without calories are allowed.

SUMMARY:
This trial examines whether 12 weeks of time-restricted eating (TRE), otherwise known as intermittent fasting, appears safe and feasible in persons with early-stage Huntington's disease (HD). The study also explores the effects of TRE on biomarkers and clinical measures associated with HD progression.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Examine the feasibility and tolerability of TRE through measures of protocol implementation, adherence rates, and adverse events.

II. Evaluate the safety of short-term TRE in the early stages of Huntington's disease (HD) by measures of body composition, vital signs, and blood analysis.

III. Analyze biomarker dynamics via peripheral markers of neurodegeneration and explore bioenergetic effects of TRE via measures of mitochondrial function.

IV. Explore whether TRE has effects on behavioral, cognitive, and motor function outcomes using standard HD clinical scales.

OUTLINE:

This study is a prospective interventional, open-label, single-arm trial. Enrolled participants are asked to engage in a TRE diet, specifically maintaining a 6-8-hour eating window every day for 12 weeks. Participants are allowed to self-select the timing of the eating window, but once selected, they are asked to maintain that schedule daily. Outside of that window, for the remaining 16-18 hours of day/night, participants are asked not to consume calorie-containing food or drink. Beverages without calories are allowed. The investigators measure body weight and composition, safety labs, adherence to the diet, dietary composition, sleep, physical activity, mood, biomarkers, and clinical outcomes. Data collection episodes take place at the Oregon Clinical and Translational Research Institute (OCTRI) within 7 days before the start of the study and again within 7 days after 12 weeks of TRE. Participants complete study surveys directly in Qualtrics.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible to participate in this study are persons who:

1. Are of at least 21 years of age at Screening.
2. Must fulfill one of the following criteria:

   1. Premanifest late prodromal HD as defined by a genetically confirmed CAG repeat greater than or equal to 36 and a CAG-Age Product (CAP) score greater than 368 (CAP = (Age) x (CAG - 33.66)).
   2. Early manifest (stage I and II) HD as defined by a TFC greater than or equal to 7. Subjects must have been determined to have a clinical diagnosis of HD by the site investigator as defined by a diagnostic confidence level (DCL) of 4.
3. Must fulfill both of the following criteria:

   1. Have undergone genetic testing with a known CAG repeat greater than or equal to 36.
   2. No features of juvenile HD (Westphal variant)

   Clarification of CAG Repeat Number (Allele length) Testing Requirements:

   A CAG repeat number obtained prior to the Screening Visit will be used to document subject eligibility if at Screening there is documentation available in the subject's record that states that the subject has an expanded CAG repeat (greater than or equal to 36) from a prior validated laboratory assessment.
4. All female subjects of childbearing potential must have a negative urine pregnancy test at baseline, and female subjects of childbearing potential must practice a highly effective method of contraception (e.g., oral contraceptives, a barrier method of birth control [e.g. condoms with contraceptive foams, diaphragms with contraceptive jelly], intrauterine devices, partner with vasectomy or sexual abstinence) for the duration of the study.
5. Are willing and capable of providing informed consent for study participation.
6. Are capable of reading, writing, and communicating effectively with others.

Exclusion Criteria:

Subjects ineligible to participate in this study are persons who:

1. Have participated in an investigational drug or device study within 30 days of the baseline visit
2. Have had previous neurosurgery for Huntington's disease or other movement disorders.
3. Have clinically significant cognitive impairment that hinders the ability to appropriately consent or adhere to detailed study directions, in the opinion of the principal investigator.
4. Have a presence of clinically significant psychosis and/or confusional states, in the opinion of the principal investigator.
5. Have clinically relevant hematologic, hepatic, cardiac, thyroid, or renal disease.
6. Have a history of substance abuse (based on DSMIV criteria) within the past 12 months prior to screening.
7. If female, are pregnant or breastfeeding.
8. Have a high-risk for nutritional deficiency.
9. Are not weight stable for at least three months prior to enrolling in the study, defined as greater than 2 kg change in body mass.
10. Express a desire to lose weight during the study.
11. Have a clinically significant medical, surgical, laboratory, or behavioral abnormality which in the judgment of the site Investigator makes the subject unsuitable for the study.
12. Have consistently practiced a time-restricted eating protocol within 3 months of trial onset.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Adherence to the TRE diet. | Week 1 to Week 13
  Adherence, measured as the number of days participants can successfully limit the eating window to 6-8 hours as tracked through self-reported surveys and time-stamped meal logs, is calculated for each participant during the 12 weeks of TRE.

SECONDARY OUTCOMES:
Change from baseline in fat-free body mass. | Baseline, Week 13
  Using bioelectrical impedance analysis, body composition, and specifically, fat-free mass (lean body mass), is measured before and after the TRE intervention.
Change from baseline in the daily eating period. | Baseline, Week 13
  The time period that participants consume calories within (from first consumption to last in the 24-hour day) is measured through retrospective survey analysis and during the lead-in week prior to the time-restricted eating (TRE) intervention. This is compared to the duration of the eating period during the 12 weeks of TRE, where participants are asked to limit the period to only 6-8 hours, while fasting the remainder of the 24 hour day.
Change from baseline in plasma neurofilament light protein (NfL). | Baseline, Week 13
  NfL is a marker of neurodegeneration and can be detected peripherally in the blood. Levels of NfL are measured before and after the TRE intervention.
Change from baseline in plasma glial fibrillary acidic protein (GFAP). | Baseline, Week 13
  GFAP is a marker of neurodegeneration and can be detected peripherally in the blood. Levels of GFAP are measured before and after the TRE intervention.
Change from baseline in the Composite Unified Huntington's Disease Rating Scale (cUHDRS). | Baseline, Week 13
  cUHDRS includes the Total Functional Capacity (range, 0-13; higher score means better functioning), Total Motor Score (range, 0-124; higher score means worse motor severity), Symbol Digit Modality Test (range, 0-110, correctly paired numbers-symbols in 90 seconds; higher score means better cognitive performance), and Stroop Word Reading (range, 0-no max value, correctly read color words in 45 seconds; higher score means better cognitive performance) scores. A z-score for each test is calculated, which alone can be used to describe relationship between an individual's test score and the mean score of a target population.

OTHER OUTCOMES:
Change from baseline in comprehensive metabolic panel values. | Baseline, Week 13
  A CMP will be drawn and analyzed before and after the TRE intervention as a safety measure.
Change from baseline in complete blood count values. | Baseline, Week 13
  A CBC will be drawn and analyzed before and after the TRE intervention as a safety measure.
Change from baseline in lipid panel values. | Baseline, Week 13
  A lipid panel will be drawn and analyzed before and after the TRE intervention as a safety measure.
Change from baseline in hemoglobin A1c. | Baseline, Week 13
  Hemoglobin A1c will be analyzed before and after the TRE intervention as a safety measure.
Change from baseline in creatinine clearance. | Baseline, Week 13
  Creatinine clearance will be analyzed before and after the TRE intervention as a safety measure.
Change from baseline in body weight. | Baseline - Week 13
  Participants are asked to self-report their body weight in a weekly survey. Every other week during the study, participants are contacted by telephone to discuss any at-home body weight changes.
Evaluation of dietary composition | Baseline - Week 13
  Twice per week, and each day during the lead-in period, participants are asked to use the SnapCalorie phone application to capture the meals eaten in a given day. Using the application, participants are asked to take photos of each meal, manually log foods, and report estimated serving sizes. Results are used to estimate caloric intake, and daily consumed fats, carbohydrates, and proteins.
Evaluation of sleep | Baseline - Week 13
  In a daily survey, participants are asked to self-report sleep duration. In a weekly survey, participants are asked to complete the Epworth Sleepiness Scale questionnaire.
Evaluation of mood | Baseline - Week 13
  In a weekly survey, participants are asked to self-report various aspects of their mood.
Evaluation of cognitive function | Baseline, Week 13
  The Montreal Cognitive Assessment (MoCA) is a validated test used to measure cognitive function. It is administered before and after the TRE intervention at the baseline and follow-up visits.
Evaluation of physical activity | Baseline - Week 13
  In a weekly survey, participants are asked to self-report the amount and type of exercise they engaged in during the previous seven days.
Evaluation of mitochondrial function | Baseline, Week 13
  Using cryopreserved peripheral blood mononuclear cells (PBMCs) isolated from participant whole blood samples drawn at the baseline and follow-up visits, mitochondrial function and electron transport chain activity are assessed with the SeahorseXF analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Amie Hiller, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make all IPD that underlie results in a publication available.
Supporting Information: Study Protocol, SAP
Time Frame: Starting June 2025
Access Criteria: Access granted to study team and data steward.

REFERENCES:
- [Background] Wells RG, Neilson LE, McHill AW, Hiller AL. Dietary fasting and time-restricted eating in Huntington's disease: therapeutic potential and underlying mechanisms. Transl Neurodegener. 2024 Apr 2;13(1):17. doi: 10.1186/s40035-024-00406-z. PMID 38561866
- [Derived] Wells RG, Neilson LE, McHill AW, Hiller AL. Time-restricted eating in early-stage Huntington's disease: A 12-week interventional clinical trial protocol. PLoS One. 2025 Mar 25;20(3):e0319253. doi: 10.1371/journal.pone.0319253. eCollection 2025. PMID 40131943